CLINICAL TRIAL: NCT06096883
Title: Development of Acetabular Erosion After Hemiarthroplasty: an Exploratory Retrospective Study
Brief Title: Hip Socket Erosion Study
Acronym: HIPSTER
Status: Enrolling by invitation | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Collaborators: Isala (Other); Jeroen Bosch Ziekenhuis (Other); Maxima Medical Center (Other); Noordwest Ziekenhuisgroep (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-2224
Record Dates: First submitted 2023-10-19; First posted 2023-10-24 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Femoral Neck Fractures; Hemiarthroplasty; Acetabulum; Protrusion
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this exploratory retrospective study is to gain a better understanding about the occurrence of acetabular erosion in patients after after hip hemiarthroplasty. The main objectives are i) to summarise a selection of basic patient characteristics of all patients of ≤ 75 years of age with a femoral neck fracture who have received either HA or THA, ii) to explore the proportion of patients after HA who developed acetabular erosion in the first years post-surgery and iii) to explore the proportion of patients after HA for whom acetabular erosion was the main reason for conversion surgery from HA to THA. A secondary objective is to assess the observer reliability of, and explore the association between, the Baker classification grading and Köhler line measurements.

All participants approached for participation in the main phase of the study will be asked to give their written informed consent to use their patient data. Patients who are willing to participate will also be asked to complete a short paper survey to collect data that is not available from their health records.

DETAILED DESCRIPTION:
Some orthopaedic surgeons believe that relatively 'young' older patients (aged ≤ 75 years) who have sustained a femoral neck fracture should be treated with hemiarthroplasty (HA) instead of total hip arthroplasty (THA). The rationale behind this belief is that THA is more time consuming, has greater associated surgical morbidity and may increase the risk of hip dislocation and subsequent revision surgery. On the other hand, HA is believed to accelerate acetabular erosion (i.e. wear) over time, which may ultimately lead to the need for conversion surgery from HA to THA. Due to a lack of research in this area, it is unclear how often the development of acetabular erosion in patients after HA actually occurs. This makes it difficult for orthopaedic surgeons to make an informed choice between HA or THA surgery for this patient group.

This is an exploratory retrospective study using existing electronic patient data of patients adhering to the inclusion criteria of the study, i.e. patients of ≤ 75 years of age who have had HA after a femoral neck fracture.

ELIGIBILITY:
Inclusion Criteria:

* having had a displaced femoral neck fracture that was subsequently treated with hemiarthroplasty
* aged < 75 years at the time of surgery
* have at least two post-operative radiographs (with at least six weeks between them) available for acetabular erosion measurements.

Exclusion Criteria:

* patients diagnosed with rheumatoid arthritis, osteoporosis, hip dysplasia or a previous hip fracture of the ipsilateral hip.

Max Age: 76 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Hospital patients who have received hemiarthroplasty after femoral neck fracture
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with acetabular erosion | Up to 15 years after index surgery
  The proportion of patients after HA who have developed acetabular erosion in the years post-surgery.

SECONDARY OUTCOMES:
The frequency of patients who have had conversion surgeries | Up to 15 years after index surgery
  The number (frequency) of patients who have had conversion surgery after the index surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Matthijs P. Somford, MD, PhD, Principal Investigator — Stichting Rijnstate Ziekenhuis
Locations (5):
- Netherlands (5):
  - Rijnstate Hospital, Arnhem, Gelderland
  - Jeroen Bosch Hospital, Department of Orthopedics, 's-Hertogenbosch
  - Northwest Clinics, Centre for Orthopaedic Research Alkmaar (CORAL) and Department of Orthopaedic Surgery, Alkmaar
  - Máxima Medical Center, Department of Orthopaedic Surgery, Eindhoven
  - Isala Hospital, Department of Orthopaedics, Zwolle

IPD SHARING:
Plan to Share IPD: Undecided